CLINICAL TRIAL: NCT05546892
Title: Short-term Outcomes of Full Bowel Preparation (MBP+OA) for Colon Resections for Cancer Versus no Bowel Preparation
Brief Title: Short-term Outcomes of Full Bowel Preparation (MBP+OA) for Colon Cancer Resections Versus no Bowel Preparation
Acronym: COLRABI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: N.N. Petrov National Medical Research Center of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COL-2
Record Dates: First submitted 2022-09-15; First posted 2022-09-21 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Colon Cancer
Keywords: colon cancer; MBP; bowel preparation; oral antibiotics
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Full bowel preparation (MBP+OA) (Experimental): Rifaximin 400 mg twice daily for three days prior to surgery
  Day prior to surgery:
  17.00 - 18.00 Macrogol-3350 - 100 g Natrium sulfate - 7,5 g Natrium chloride - 2,691 g Potassium chloride - 1,015 g Ascorbic acid - 4,7 g Natrii ascorbate - 5,9 g Clear fluids - 1000 ml
  18.00 - 19.00 Clear fluids 500 ml
  19.00 - 20.00 Macrogol-3350 - 100 g Natrium sulfate - 7,5 g Natrium chloride - 2,691 g Potassium chloride - 1,015 g Ascorbic acid - 4,7 g Natrii ascorbate - 5,9 g Clear fluids - 1000 ml
  20.00 - 21.00 Clear fluids 500 ml
  Interventions: Procedure: Full bowel preparation prior to colon resection for cancer
- No bowel preparation (Active Comparator): No bowel preparation (enema of not more then 500 ml is allowed prior or during surgery)
  Interventions: Procedure: No bowel preparation

INTERVENTIONS:
Procedure: Full bowel preparation prior to colon resection for cancer — Mechanical bowel preparation and oral antibiotics
  Arms: Full bowel preparation (MBP+OA)
Procedure: No bowel preparation — Omission of any bowel preparation
  Arms: No bowel preparation

SUMMARY:
The purpose of the study is to determine if short-term outcomes of colon resections after full bowel preparation (mechanical bowel preparation plus oral antibiotics) are superior to colon resections with no bowel preparation.

DETAILED DESCRIPTION:
The design involves random allocation of eligible patients to full bowel preparation or no bowel preparation in 1:1 ratio. After that colon resection is performed in both groups.

Short-term outcomes are assessed in 30 day period after surgery. This is a superiority trial evaluating statistical superiority. Rate of anastomotic leak is anticipated to decrease from 8% (data from local registry) to 3%. For power of 80% enrolment of 586 patients is required.

The intent-to-treat principle is used for the data analysis.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed adenocarcinoma of the colon (caecum, ascending, transverse, descending, sigmoid)
* clinical stage T1-4aN0-2M0-1 (distant metastases must be resectable)
* indications for surgical colonic resection
* ECOG status 0-2
* At least 18 years of age
* Written informed consent

Exclusion Criteria:

* Medical or psychiatric conditions that compromise the patient's ability to give informed consent or comply with the study protocol
* Pregnancy or breast feeding
* Medical contraindications for surgical treatment
* Any use of antibiotics 30 days prior to inclusion
* Functioning stoma
* Contraindications for use of MBP or OA drugs or their components
* Indications for mandatory MBP (planned intraoperative colonoscopy etc)
* Indications for obstructive resection
* Acute bowel obstruction, bleeding or perforation
* Other malignancies not in remission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 586 (Estimated)
Dates: Start 2023-02-10 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Anastomotic leak rate | 30 days
  Rate of anastomotic leak in patients after colon resections

SECONDARY OUTCOMES:
Surgical site infection (SSI) rate | 30 days
  Rate of Surgical site infection
Intraabdominal and or pelvic abscess rate | 30 days
  Rate of intraabdominal and or pelvic abscess
Overall morbidity | 30 days
  Rate of patients with any complications after surgery
Rate of intraoperative complications | Duration of surgical procedure
  Rate of patients with intraoperative complications
Surgery duration in minutes | Duration of surgical procedure
  Time of surgical procedure
Quality of bowel preparation assessed by surgeon | Day of surgical procedure
  Assessment of bowel preparation quality by surgeon (qualitative scale)
Bowel preparation compliance | Day of surgical procedure
  Rate of patients in experimental arm undergoing complete bowel preparation according to protocol

CONTACTS AND LOCATIONS:
Overall Officials: Aleksei Karachun, Study Chair — N.N. Petrov National Medical Research Center of Oncology
Locations (1):
- N.N. Petrov National Medical Research Center of Oncology, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No
We are not planning to share individual participant data